CLINICAL TRIAL: NCT01319370
Title: Investigator-Initiated, Double Blind, Two-Armed, Placebo-Controlled, Randomized Clinical Trial With an Open-Label Extension Phase, to Investigate Efficacy of 5% Minoxidil Topical Foam Twice Daily in Men With Androgenetic Alopecia in the Temple and Vertex Region Concerning Hair Volume Over 24 / 104 Weeks
Brief Title: Effectiveness and Safety of Minoxidil Foam Versus Placebo Foam for Androgenetic Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Natalie GARCIA BARTELS (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, Natalie GARCIA BARTELS, PD, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRC-AGA02; 2010-018291-25 (EudraCT Number)
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vehicle of 5% Minoxidl topical foam (Placebo Comparator): vehicel foam in twice daily application in temple and vertex region
  Interventions: Drug: vehicle of 5% Minoxidil topical foam
- 5% Minoxidil topical foam (Active Comparator): 5% Minoxidil topical in twice daily application in temple and vertex region
  Interventions: Drug: Minoxidil

INTERVENTIONS:
Drug: Minoxidil — 1 g of 5% Minoxidil topical foam twice daily over 24 weeks in double-blinded phase and further 80 weeks in open-label-phase
  Arms: 5% Minoxidil topical foam
Drug: vehicle of 5% Minoxidil topical foam — 1 g of vehicle topical foam twice daily over 24 weeks in double-blinded phase and further 80 weeks in open-label-phase
  Arms: vehicle of 5% Minoxidl topical foam

SUMMARY:
The current study aims to show efficacy of twice daily application of 5% Minoxidil Topical Foam (MTF) formulation compared to placebo in the temple region of male patients with androgenetic alopecia after 24 weeks as well as to gain long-term data on the efficacy and safety of 5% MTF in male subjects with AGA in temple and vertex region, over a period of 2 years. Objective and subjective efficacy measures will be compared to baseline. Moreover, all patients will get the equal treatment and measurements in the vertex region to enable comparison of the efficacy of 5% Minoxidil Topical Foam in the temples not only to baseline but also to vertex region. Additionally safety assessments will be performed throughout the whole study.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18 to 70 year old, in general good health
* Exhibits male AGA based on a discernable hair loss in temple and vertex region rating Hamilton-Norwood Scale III vertex to VI (See Appendix 1)
* Subjects who give their consent to the study after thorough explanation and who personally signed and dated the informed consent document indicating that the subject, has been informed of all pertinent aspects of the trial
* Willing to maintain the same hairstyle, hair length and hair color throughout the study
* Subjects who are willing and able to comply with scheduled visits, treatment plan, mini-tattoo and other trial procedures
* Accepting the Information form plus accepting and signing the Informed Consent form

Exclusion Criteria:

* Known to be hypersensitive to minoxidil, hair dye (p-phenylenediamine), tattoo ink, fragrances, hair gel or any vehicle components
* Current or 4 weeks dated back use of medical shampoos or solutions which include Ketoconazole or the like (e. g. Terzolin®) in the target region interfering with the CTM or examination method
* Current or 3 months dated back use of topical treatment in the target regions taken for more then 2 consecutive weeks interfering with the CTM (topical corticosteroids, aminexil, minoxidil, estrogens)
* Current or 3 months dated back use of systemic treatment (drugs or dietary supplement) taken for more than 2 consecutive weeks interfering with the CTM or examination method (beta blocker, cimetidine, diazoxide, isotretionin, corticosteroids, vitamin A intake above 10000 IU per day)
* Current or 12 months dated back use of Finasteride (Propecia®, FinaHair®, etc.), Dutasteride or a similar product
* Within past 12 months undergoing chemotherapy or receiving cytotoxic agents as well as radiation and/or laser/surgical therapy of the scalp
* Current or prior enrollment in any other investigational medication (drug) study within the 4 weeks prior to study initiation
* Presence of hair transplants, hair weaves or non-breathable wigs and hair bonding
* Current or 2 months dated back severe diet or presenting a history of eating disorder
* Any dermatological disorders of the scalp in the target region with the possibility of interfering with the CTM or examination method, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars or scalp atrophy
* Untreated persisting hypertension
* Active hair loss or history within the past 3 months including diffuse telogen effluvium, alopecia areata, scarring alopecia
* Other severe, acute or chronic medical condition that may lead to hair loss or interfere with the interpretation of trial results (e. g. untreated hypothyroidism)
* Individuals who are institutionalized by court or regulatory order

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change of target area non-vellus hair count in the temple region (t-TAHC) [n/cm²] compared to baseline after 24 weeks | Baseline, week 8, week 16, week 24, week 52, week 76, week 104

SECONDARY OUTCOMES:
Assessing the investigational products safety by means of clinical examination (local intolerance, AE, SAE) | every visit from baseline to week 104
Change of cumulative hair width in non-vellus hair in temple and vertex region (t-TAHW; v-TAHW) [mm/cm²] compared to baseline after 24, 52, 76 and 104 weeks | Baseline, week 8, week 16, week 24, week 52, week 76, week 104
Change of t-TAHC, v-TAHC, t-TAHW and v-TAHW comparing 5% MTF and Placebo Topical Foam (plaTF) groups | Baseline, week 8, week 16, week 24, week 52, week 76, week 104
Global expert panel and subjects' rating change in scalp coverage: week 24 compared to baseline, week 104 compared to baseline and week 104 compared to week 24 via assessment of global temple and vertex photographs | Baseline, week 8, week 16, week 24, week 52, week 76, week 104

CONTACTS AND LOCATIONS:
Locations (1):
- Charité-Universitätsmedizin Berlin, Clinical Research Center for Hair and Skin Science, Dept. of Dermatology, Venereology and Allergy, Berlin, Germany